CLINICAL TRIAL: NCT03391284
Title: Preemptive Oral vs Intravenous Acetominophen for Postoperative Pain in Minimally Invasive Gynecologic Surgery: A Randomized Control Trial
Brief Title: Oral vs Intravenous Acetominophen for Postoperative Pain in Minimally Invasive Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Bruce Kahn, PI, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCRIPPS-WHR-ACET-01
Record Dates: First submitted 2016-01-09; First posted 2018-01-05 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Acetominophen Arm (Experimental): 1000 mg acetominophen oral
  Interventions: Drug: acetominophen; Drug: Acetaminophen
- Intravenous (Active Comparator): 1000 mg acetominophen intravenous
  Interventions: Drug: acetominophen; Drug: Acetaminophen

INTERVENTIONS:
Drug: acetominophen — INTRAVENOUS
  Other Names: Ofirmev
Drug: Acetaminophen — ORAL
  Other Names: Tylenol

SUMMARY:
Hypothesis: Postoperative pain will be equivalent in patients receiving preemptive oral acetaminophen as compared to patients receiving preemptive intravenous acetaminophen following minimally invasive benign gynecologic surgery.

Primary outcome:

• Difference in postoperative pain comparing preemptive use of PO versus IV acetaminophen

o Mean Visual analog Scale (VAS) scores will be compared between the intervention group (PO acetaminophen) and the control group (IV acetaminophen).

Secondary outcomes:

* Difference in postoperative analgesic use between groups

  o Narcotics, NSAIDs
* Difference in postoperative N/V between groups

  o Patient rated measure - none, mild, moderate, severe
* Cost comparison between drugs

DETAILED DESCRIPTION:
Hypothesis: Postoperative pain will be equivalent in patients receiving preemptive oral acetaminophen as compared to patients receiving preemptive intravenous acetaminophen following minimally invasive benign gynecologic surgery.

Importance/significance: Adequate control of postoperative pain is important for patient satisfaction, adequate healing, and optimizing length of stay. The idea of preemptive analgesia (giving an analgesic prior to first skin incision to prevent sensitization of nerve pathways from the trauma of surgery) has been shown in many studies to improve postoperative pain. Intravenous acetaminophen has been found to be an effective agent when given preemptively, and many surgeons have adopted this practice. Unfortunately, the IV formulation of acetaminophen, unlike the oral formulation, is expensive as it is a relatively new drug. There are other oral analgesics (i.e. Celebrex) that have been found to be efficacious for postoperative pain control when given preemptively. There are no studies in gynecologic surgery, however, comparing the effectiveness of PO acetaminophen with IV acetaminophen. Given that PO acetaminophen is significantly cheaper than the IV formulation, this could result in cost savings for hospital systems while maintaining adequate patient comfort and satisfaction.

Primary outcome:

1. Difference in postoperative pain comparing preemptive use of PO versus IV acetaminophen
2. Mean VAS scores will be compared between the intervention group (PO acetaminophen) and the control group (IV acetaminophen).

Secondary outcomes:

1. Difference in postoperative analgesic use between groups - Narcotics, NSAIDs
2. Difference in postoperative N/V between groups
3. Patient rated measure - none, mild, moderate, severe
4. Cost comparison between drugs

Methods:

Patients scheduled to undergo minimally invasive benign gynecologic surgery will be randomized to one of two groups:

Group 1: acetaminophen 1 gram PO 30min before surgery, then saline placebo IV after anesthesia induction but before skin incision

Group 2: receives placebo pill PO 30min before surgery, then acetaminophen 1 gram IV after anesthesia induction but before skin incision

Primary outcome: After surgery, postoperative pain measured at various time points by blinded investigator

2 hours postop, 4 hours postop, 24 hours postop

Secondary outcomes:

1. Evaluate N/V - self-rated as none, mild, moderate, severe
2. Document amount of analgesic use (narcotic, NSAIDs) during hospital course
3. Compute cost comparison between medications

Demographics to collect:

Age, parity, BMI, procedure indication, pathology including uterine weight, procedure length

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older scheduled to undergo robotic-assisted laparoscopic hysterectomy for benign conditions.

Exclusion Criteria:

* Known or suspected malignancy,
* Active liver/renal disease,
* Chronic alcohol use/alcoholism,
* Allergy to acetaminophen,
* Conversion to laparotomy,
* hx gastroparesis,
* Poorly controlled insulin dependent diabetes or gastric bypass surgery,
* Regular/recent (past 6 months) narcotic use,
* Inability to swallow pills.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Pain - VAS | 2 hours
  Pain level 2 hours post treatment

SECONDARY OUTCOMES:
Pain - VAS | 4 hours
  Pain level 4 hours post treatment
Pain - VAS | 24 hours
  Pain level 24 hours post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Kahn, MD, Principal Investigator — Scripps
Locations (2):
- United States (2):
  - Scripps Clinic, San Diego, California
  - Scripps Clininc Dept of Ob/Gyn, San Diego, California

REFERENCES:
- [Derived] Lombardi TM, Kahn BS, Tsai LJ, Waalen JM, Wachi N. Preemptive Oral Compared With Intravenous Acetaminophen for Postoperative Pain After Robotic-Assisted Laparoscopic Hysterectomy: A Randomized Controlled Trial. Obstet Gynecol. 2019 Dec;134(6):1293-1297. doi: 10.1097/AOG.0000000000003578. PMID 31764741